CLINICAL TRIAL: NCT01294683
Title: A Phase III Multicenter, Double-Blind, Crossover Design Study to Evaluate Lipid-Altering Efficacy and Safety of Extended-Release Niacin/Laropiprant/Simvastatin Combination Tablet in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: A Study to Evaluate Efficacy and Safety of Extended-Release Niacin + Laropiprant + Simvastatin in Participants With Primary Hypercholesterolemia or Mixed Dyslipidemia (MK-0524B-118)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0524B-118; 2010-023939-42 (EudraCT Number)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Primary Hypercholesterolemia; Dyslipidemia
Keywords: Low-density lipoprotein; LDL; High-density lipoprotein; HDL; Niacin; Lipid modifying therapy; Cholesterol; High cholesterol; Triglycerides; Mixed Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — Simvastatin; Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1: MK-0524B 2g/40g→MK-0524A 2g + Simvastatin 40 mg (Experimental): After a 2-week placebo run-in, participants received extended release (ER) niacin/laropiprant (N/LRPT) 1 g/20 mg combination tablet (MK-0524B) once daily for 4 weeks, then ERN/LRPT/Simvastatin (SIM) 2 g/40 mg combination tablet once daily for 8 weeks. Participants then received ERN/LRPT 2 g (MK-0524A) co-administered with SIM 40 mg once daily for 8 weeks.
  Interventions: Drug: Simvastatin; Drug: Extended Release (ER) niacin/laropiprant/simvastatin (N/LRPT/SIM); Drug: Extended Release (ER) niacin/laropiprant (N/LRPT); Drug: Placebo
- Sequence 2: MK-0524A 2g + Simvastatin 40 mg→ MK-0524B 2g/40g (Experimental): After a 2-week placebo run-in, participants received ERN/LRPT 1 g (MK-0524A) co-administered with SIM 20 mg once daily for 4 weeks then received ERN/LRPT 2 g (MK-0524A) co-administered with SIM 40 mg once daily for 8 weeks. Participants then received ERN/LRPT/SIM 2 g/40 mg combination tablets (MK-0524B) once daily for 8 weeks.
  Interventions: Drug: Simvastatin; Drug: Extended Release (ER) niacin/laropiprant/simvastatin (N/LRPT/SIM); Drug: Extended Release (ER) niacin/laropiprant (N/LRPT); Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin
  Other Names: Zocor
Drug: Extended Release (ER) niacin/laropiprant/simvastatin (N/LRPT/SIM)
  Other Names: MK-0524B
Drug: Extended Release (ER) niacin/laropiprant (N/LRPT)
  Other Names: MK-0524A
Drug: Placebo

SUMMARY:
This study is being done to find out if tablets containing extended release (ER) niacin, laropiprant, and simvastatin (ERN/LRPT/SIM) are as effective as tablets containing ER niacin and laropiprant taken with simvastatin tablets (ERN/LRPT + SIM) for lowering high cholesterol and high lipid levels in the blood. The primary hypothesis is that ERN/LRPT/SIM 2 g/40 mg is equivalent to ERN/LRPT 2 g co-administered with simvastatin 40 mg in reducing low-density lipoprotein cholesterol (LDL-C).

ELIGIBILITY:
Inclusion criteria

* Participant has a history of primary hypercholesterolemia or mixed dyslipidemia and meets LDL-C and triglyceride criteria.
* Visit 2:
* Participant is high risk coronary heart disease (CHD) or CHD risk-equivalent.

Exclusion Criteria

* Participant is pregnant or breast-feeding, or expecting to conceive during the study.
* Participant has a history of malignancy.
* Participant consumes more than 3 alcoholic drinks per day (14 per week).
* Participant is high risk CHD patient on statin therapy or any patient on statin therapy equivalent to 80 mg simvastatin.
* Participant with Type 1 or Type 2 diabetes mellitus that is poorly controlled, or on statin therapy.
* Participant currently engages in vigorous exercise or is on an aggressive diet regimen.
* Participant uncontrolled endocrine or metabolic disease, uncontrolled gout, kidney or hepatic disease, heart failure, recent peptic ulcer disease, hypersensitivity or allergic reaction to niacin or simvastatin, recent heart attack, stroke or heart surgery.
* Participant is human immunodeficiency virus (HIV) positive.
* Participant has taken niacin >50 mg/day, bile-acid sequestrants, hydroxymethyl glutaryl coenzyme A (HMG-CoA) reductase inhibitors, ezetimibe, Cholestin™ [red yeast rice] and other red yeast products within 6 weeks, or fibrates within 8 weeks of randomization visit (Visit 3).

  * Note: Fish oils, phytosterol margarines and other non-prescribed therapies are allowed provided participant has been on a stable dose for 6 weeks prior to Visit 2 and agrees to remain on this dose for the duration of the study.
* Participant is currently receiving cyclical hormonal contraceptives or intermittent use of hormone replacement therapies (HRTs) (e.g., estradiol, medroxyprogesterone, progesterone).

  * Note: Participants who have been on a stable dose of non-cyclical HRT or hormonal contraceptive for greater than 6 weeks prior to Visit 1 are eligible if they agree to remain on the same regimen for the duration of the study.
* Participant is taking prohibited medications such as systemic corticosteroids, itraconazole or ketoconazole, erythromycin, clarithromycin, or telithromycin, nefazodone, HIV protease inhibitors, verapamil, amiodarone, cyclosporine, danazol, diltiazem or fusidic acid.
* Participant consumes >1 quart of grapefruit juice/day.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 977 (Actual)
Dates: Start 2011-02-04 (Actual); Primary Completion 2012-01-17 (Actual); Study Completion 2012-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/study.html?id=0524B-118&kw=0524B-118&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a 6-8 week washout then completed a 2-week placebo run-in prior to the start of active treatment.
Groups:
- Sequence 1: MK-0524B 2g/40g→MK-0524A 2g + Simvastatin 40 mg: After a 2-week placebo run-in, participants received extended release niacin/laropiprant (ERN/LRPT) 1 g/20 mg combination tablet (MK-0524B) once daily for 4 weeks, then ERN/LRPT/Simvastatin (SIM) 2 g/40 mg combination tablet once daily for 8 weeks. Participants then received ERN/LRPT 2 g (MK-0524A) co-administered with SIM 40 mg once daily for 8 weeks.
Period: Precrossover (Periods I/II)
Arm/Group | Sequence 1: MK-0524B 2g/40g→MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524A 2g + Simvastatin 40 mg→ MK-0524B 2g/40g
Started | 489 | 488
Treated | 486 | 486
Completed | 232 | 222
Not Completed | 257 | 266
Not completed — Adverse Event | 49 | 52
Not completed — Lost to Follow-up | 3 | 6
Not completed — Non-compliance with Study Drug | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 5 | 5
Not completed — Study Terminated by Sponsor | 187 | 192
Not completed — Technical Problems | 0 | 1
Not completed — Withdrawal by Subject | 11 | 9
Period: Post Crossover (Period III)
Arm/Group | Sequence 1: MK-0524B 2g/40g→MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524A 2g + Simvastatin 40 mg→ MK-0524B 2g/40g
Started | 232 | 222
Completed | 199 | 190
Not Completed | 33 | 32
Not completed — Adverse Event | 6 | 6
Not completed — Lost to Follow-up | 1 | 3
Not completed — Study Terminated by Sponsor | 23 | 21
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: MK-0524B 2g/40g→MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524A 2g + Simvastatin 40 mg→ MK-0524B 2g/40g | Total
Number analyzed (Participants) | 489 | 488 | 977
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.2) | 57.9 (10.2) | 56.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 258 | 488
  Male | 259 | 230 | 489

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Blood samples were taken at baseline (Week 4 for Period II; Week 12 for Period III) and after 8 weeks of treatment (Week 12 for Period II and Week 20 for Period III) to determine the LDL-C levels. The change from baseline after 8 weeks of treatment was recorded.
  Results from recent studies indicated that the combination tablet formulations used in the study did not meet the pre-specified pharmacokinetic bounds used to establish the equivalence of the combination tablet (MK-0524B; ERN/LRPT/SIM) to the coadministration of MK-0524A (ERN/LRPT) and SIM. Therefore, efficacy data were not analyzed, as the study was stopped early. Only safety data were evaluated.
Time Frame: Baseline (Week 4 for Period II; Week 12 for Period III) and after 8 weeks of treatment (Week 12 for Period II and Week 20 for Period III)
Population: Study was terminated by the Sponsor prior to completion. No planned efficacy summaries or analyses were completed.
Groups:
- MK-0524B 2g/40mg: Participants who received MK-0524B 2g/40mg for 8 weeks in either Period II or Period III regardless of randomly assigned sequence.
- MK-0524A 2g + Simvastatin 40 mg: Participants who received MK-0524A 2g+Simvastatin 40mg for 8 weeks in either Period II or Period III regardless of randomly assigned sequence.
Arm/Group | MK-0524B 2g/40mg | MK-0524A 2g + Simvastatin 40 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C)
Description: Blood samples were taken at baseline (Week 4 for Period II; Week 12 for Period III) and after 8 weeks of treatment (Week 12 for Period II and Week 20 for Period III) to determine the HDL-C levels. The change from baseline after 8 weeks of treatment was recorded.
  Results from recent studies indicated that the combination tablet formulations used in the study did not meet the pre-specified pharmacokinetic bounds used to establish the equivalence of the combination tablet (MK-0524B; ERN/LRPT/SIM) to the coadministration of MK-0524A (ERN/LRPT) and SIM. Therefore, efficacy data were not analyzed, as the study was stopped early. Only safety data were evaluated.
Time Frame: Baseline (Week 4 for Period II; Week 12 for Period III) and after 8 weeks of treatment during each period (Week 12 for Period II and Week 20 for Period III)
Population: Study was terminated by the Sponsor prior to completion. No planned efficacy summaries or analyses were completed.
Arm/Group | MK-0524B 2g/40mg | MK-0524A 2g + Simvastatin 40 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Consecutive Elevations in Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) of >=3 x Upper Limit of Normal (ULN)
Description: Participants had AST and ALT levels assessed during Period I (4 weeks ) and throughout each 8 week treatment period (20 weeks total). Participants who had an assessment of either AST or ALT that was 3 x ULN or greater were recorded. The AST UNLs for males and females were 43 U/L and 36 U/L, respectively. The ALT UNLs for males and females were 40 U/L and 33 U/L, respectively.
Time Frame: Up 20 weeks (12 weeks in Periods I/II and 8 weeks in Period III)
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 postbaseline measurement within 14 days of the last dose of study drug. Analysis was based on the experiences accumulated during Periods I/II combined, where the study followed a parallel design. A separate safety analysis was performed for Period III.
Measure: Number; unit: Percentage of Participants
Groups:
- Sequence 1: MK-0524B 2g/40g: Participants who received MK-0524B 1g/40mg and MK-0524B 2g/40mg during Periods I/II
- Sequence 2: MK-0524A 2g + Simvastatin 40 mg: Participants who received MK-0524A 1g + Simvastatin 40mg and MK-0524A 2g+ Simvastatin 40mg during Periods I/II.
- Sequence 1: MK-0524A 2g + Simvastatin 40 mg: Participants who received MK-0524A 2g+ Simvastatin 40mg during Period III.
- Sequence 2: MK-0524B 2g/40g: Participants who received MK-0524B 2g/40mg during Period III
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 0.4 | 0.6 | 1.3 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 2g/40g vs Sequence 2: MK-0524A 2g + Simvastatin 40 mg; Periods I/II; Test type: Superiority or Other; p = 0.654, Miettinen and Nurminen; Difference in Percentages = -0.206, 95% CI 2-sided [-1.434 to 0.936]
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g + Simvastatin 40 mg vs Sequence 2: MK-0524B 2g/40g; Period III; Test type: Superiority or Other; p = 0.090, Miettinen and Nurminen; Difference in Percentages = 1.304, 95% CI 2-sided [-0.427 to 3.768]

4. Secondary Outcome: Percentage of Participants With Elevations in ALT and/or AST of >=5 x ULN
Description: Participants had AST and ALT levels assessed during Period I (4 weeks ) throughout each 8 week treatment period (20 weeks total). Participants who had an assessment of either AST or ALT that was 5 x ULN or greater were recorded. The AST UNLs for males and females were 43 U/L and 36 U/L, respectively. The ALT UNLs for males and females were 40 U/L and 33 U/L, respectively.
Time Frame: up 20 weeks (12 weeks in Periods I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 0.2 | 0.4 | 0.9 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 2g/40g vs Sequence 2: MK-0524A 2g + Simvastatin 40 mg; Periods I/II; Test type: Superiority or Other; p = 0.563, Miettinen and Nurminen; Difference in Percentages = -.206, 95% CI 2-sided [-1.303 to 0.779]
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g + Simvastatin 40 mg vs Sequence 2: MK-0524B 2g/40g; Period III; Test type: Superiority or Other; p = 0.166, Miettinen and Nurminen; Difference in Percentages = 0.870, 95% CI 2-sided [-0.858 to 3.118]

5. Secondary Outcome: Percentage of Participants With Elevations in ALT and/or AST of >=10 x ULN
Description: Participants had AST and ALT levels assessed during Period I (4 weeks ) throughout each 8 week treatment period (20 weeks total). Participants who had an assessment of either AST or ALT that was 10 x ULN or greater were recorded. The AST UNLs for males and females were 43 U/L and 36 U/L, respectively. The ALT UNLs for males and females were 40 U/L and 33 U/L, respectively.
Time Frame: up 20 weeks (12 weeks in Periods I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0

6. Secondary Outcome: Percentage of Participants With Creatine Kinase (CK) >=10 x ULN
Description: Participants had CK levels assessed throughout the treatment periods. Participants who had any CK level that was >=10 x ULN were recorded. The UNLs for males and females were 207 U/L and 169 U/L, respectively.
Time Frame: up 20 weeks (12 weeks in Periods I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 0.0 | 0.0 | 0.9 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524A 2g + Simvastatin 40 mg vs Sequence 2: MK-0524B 2g/40g; Period III; Test type: Superiority or Other; p = 0.166, Miettinen and Nurminen; Difference in Percentages = 0.870, 95% CI 2-sided [-0.858 to 3.118]

7. Secondary Outcome: Percentage of Participants With CK >=10 x ULN With Muscle Symptoms - Drug Related
Description: Participants had CK levels assessed throughout the treatment periods. Participants who had any CK level that was >=10 x ULN and had associated muscle symptoms present within +/- 7 days that were reported as at least possibly related to study drug were recorded. The UNLs for males and females were 207 U/L and 169 U/L, respectively.
Time Frame: up 20 weeks (12 weeks in Periods I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants Who Experienced at Least 1 Hepatitis-related Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. Hepatitis-related AEs were identified by a collective review using the following pre-specified set of preferred terms: cholestasis, hepatic necrosis, hepatocellular damage, cytolytic hepatitis, hepatitis, hepatomegaly, jaundice, hepatic failure, hepatitis cholestatic, jaundice cholestatic, hepatitis fulminant, hyperbilirubinaemia, jaundice hepatocellular, ocular icterus, yellow skin, hepatic function abnormal, acute hepatic failure, subacute hepatic failure, hepatitis acute, hepatitis toxic, hepatotoxicity, and mixed hepatocellular-cholestatic injury.
Time Frame: up 20 weeks (12 weeks in Periods I/II and 8 weeks in Period III)
Population: All participants who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined (pre-crossover), where the study followed a parallel design. A separate safety analysis was performed for Period III (post-crossover).
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0

9. Secondary Outcome: Percentage of Participants With New Onset of Diabetes
Description: Participants who with newly diagnosed of diabetes were recorded. A participant was classified as having new onset diabetes if they experienced an AE related to a diagnosis of diabetes (based on a pre-defined set of Medical Dictionary for Regulatory Activities [MedDRA] terms), or if they started taking an anti-diabetic medication during the course of the study. The MedDRA terms were as follows: diabetes mellitus, diabetes mellitus insulin-dependent, diabetes mellitus non-insulin dependent, insulin-requiring type II diabetes mellitus, insulin resistant diabetes, diabetes with hyperosmolarity, latent autoimmune diabetes in adults.
Time Frame: up 20 weeks (12 weeks in Periods I/II and 8 weeks in Period III)
Population: All participants without diabetes at baseline and who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined (pre-crossover), where the study followed a parallel design. A separate safety analysis was performed for Period III (post-crossover).
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 1.0 | 0.4 | 1.3 | 0.9
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 2g/40g vs Sequence 2: MK-0524A 2g + Simvastatin 40 mg; Periods I/II; Test type: Superiority or Other; p = 0.255, Miettinen and Nurminen; Difference in Percentages = 0.617, 95% CI 2-sided [-0.575 to 2.023]
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g + Simvastatin 40 mg vs Sequence 2: MK-0524B 2g/40g; Period III; Test type: Superiority or Other; p = 0.690, Miettinen and Nurminen; Difference in Percentages = 0.395, 95% CI 2-sided [-2.091 to 2.966]

10. Secondary Outcome: Percentage of Participants With a Confirmed Adjudicated Cardiovascular Event
Description: Select serious adverse cardiovascular events and all-cause mortality that occurred during the treatment phase of the study were adjudicated by an expert committee external to the sponsor. Those events confirmed by the committee a cardiovascular events were recorded.
Time Frame: up 20 weeks (12 weeks in Periods I/II and 8 weeks in Period III)
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 0.2 | 0.2 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 2g/40g vs Sequence 2: MK-0524A 2g + Simvastatin 40 mg; Periods I/II; Test type: Superiority or Other; p > 0.999, Miettinen and Nurminen; Difference in Percentages = 0.000, 95% CI 2-sided [-0.967 to 0.967]

11. Secondary Outcome: Percentage of Participants Who Experienced at Least 1 AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE.
Time Frame: up 22 weeks (12 weeks in Periods I/II and 10 weeks in Period III)
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 50.2 | 51.2 | 30.4 | 29.5
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 2g/40g vs Sequence 2: MK-0524A 2g + Simvastatin 40 mg; Periods I/II; Test type: Superiority or Other; Miettinen and Nurminen; Difference in Percentages = -1.029, 95% CI 2-sided [-7.301 to 5.252] — Miettinen and Nurminen Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g + Simvastatin 40 mg vs Sequence 2: MK-0524B 2g/40g; Period III; Test type: Superiority or Other; Difference in Percentages = 0.889, 95% CI 2-sided [-7.599 to 9.338] — Miettinen and Nurminen Method

12. Secondary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. Participants who were discontinued from the study due to an AE were recorded.
Time Frame: up 22 weeks (12 weeks in Periods I/II and 10 weeks in Period III)
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Number analyzed (Participants) | 486 | 486 | 230 | 220
Percentage of Participants | 10.1 | 10.5 | 2.2 | 2.7
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 2g/40g vs Sequence 2: MK-0524A 2g + Simvastatin 40 mg; Periods I/II; Test type: Superiority or Other; Difference in Percentages = -0.412, 95% CI 2-sided [-4.280 to 3.450]
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g + Simvastatin 40 mg vs Sequence 2: MK-0524B 2g/40g; Period III; Test type: Superiority or Other; Difference in Percentages = -0.533, 95% CI 2-sided [-3.916 to 2.619] — Miettinen and Nurminen Method

ADVERSE EVENTS:
Time Frame: up 22 weeks (12 weeks in Periods I/II and 10 weeks in Period III)
Description: Population included all participants who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined (pre-crossover), where the study follows a parallel design. A separate safety analysis was performed for Period III (post-crossover).
Arm/Group | Sequence 1: MK-0524B 2g/40g | Sequence 2: MK-0524A 2g + Simvastatin 40 mg | Sequence 1: MK-0524A 2g + Simvastatin 40 mg | Sequence 2: MK-0524B 2g/40g
Serious Adverse Events (participants affected / at risk) | 6/486 | 9/486 | 1/230 | 5/220
Other Adverse Events (participants affected / at risk) | 110/486 | 98/486 | 0/230 | 0/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sequence 1: MK-0524B 2g/40g (N=486) | Sequence 2: MK-0524A 2g + Simvastatin 40 mg (N=486) | Sequence 1: MK-0524A 2g + Simvastatin 40 mg (N=230) | Sequence 2: MK-0524B 2g/40g (N=220)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1: MK-0524B 2g/40g (N=486) | Sequence 2: MK-0524A 2g + Simvastatin 40 mg (N=486) | Sequence 1: MK-0524A 2g + Simvastatin 40 mg (N=230) | Sequence 2: MK-0524B 2g/40g (N=220)
Pruritus (Skin and subcutaneous tissue disorders) | 42 (51) | 33 (38) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 88 (104) | 75 (86) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.